CLINICAL TRIAL: NCT03952260
Title: A Randomised Control Trial Comparing 6-4-1 Fasting Protocol Against Classical 6-4-2 Fasting Guideline for Paediatric Patients
Brief Title: Feasibility of 1 Hour Clear Fluid Fasting Prior to Paediatric GA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ma Tai Jiun (Other)
Responsible Party: Sponsor-Investigator, Ma Tai Jiun, Principal investigator, University of Malaya
Organization: University of Malaya (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019211-7120
Record Dates: First submitted 2019-05-04; First posted 2019-05-16 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Gastric Residual Volume
Keywords: Clear fluid fasting; residual gastric volume; paediatric anaesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded against those who are doing ultrasound assessment of gastric residual volume prior to anaesthesia
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting clear fluid for 1 hour prior to anaesthesia (Active Comparator): Fasting clear fluid for 1 hour prior to anaesthesia
  Interventions: Other: Fasting time for clear fluid prior to anaesthesia
- Fasting clear fluid for 2 hours prior to anaesthesia (No Intervention): Fasting clear fluid for 2 hours prior to anaesthesia

INTERVENTIONS:
Other: Fasting time for clear fluid prior to anaesthesia — This study is to evaluate the latest fasting protocol that is currently adopted and recommended by United Kingdom, France and Royal Children Hospital Melbourne.
  The research question is should we change our fasting protocol for paediatric patients prior to operation The anaesthesia service is being studied. Prior to induction, the amount of abdominal contents was examined using ultrasound scan. In addition, parents will complete a questionnaire after the surgery to assess anxiety level of patients before and after the surgery.
  Arms: Fasting clear fluid for 1 hour prior to anaesthesia

SUMMARY:
The study is aim to investigate the appropriate fasting time for clear fluid in paediatric patients who plan for elective minor surgery.

This is a randomize control trial, which patient will be selected randomly to fast for clear fluid for 1 hour or 2 hours.

It is important to determine the gastric residual volume for paediatric age group prior to elective minor surgery in order to determine whether the difference between 1 hour fasting and 2 hour fasting for clear fluid is significant.

DETAILED DESCRIPTION:
This study is to evaluate the latest fasting protocol that is currently adopted and recommended by United Kingdom, France and Royal Children Hospital Melbourne.

The research question is should investigator change fasting protocol for paediatric patients prior to operation.

The anaesthesia service is being studied. Participants are patients who are 5-16 years old are planned for elective minor surgery in ent, eye, dental surgery, general surgery and orthopaedics.

This study will be done in UMMC. 2 groups of patients will be recruit which consists of 50 patients each. Each of the group will be instructed to fast for clear fluid for 1 hour or 2 hours prior to surgery. Prior to induction, the amount of abdominal contents was examined using ultrasound scan. In addition, patients anxiety level prior to and 1 hour post general anaesthesia will be assess. Also, parents of patients will complete a questionnaire after the surgery to assess parental satisfaction toward anaesthesia service.

ELIGIBILITY:
Inclusion Criteria:

* 5-16 years old
* elective open minor surgery in ent, eye, dental surgery, general surgery and orthopaedics

Exclusion Criteria:

* Gastro-oesophageal reflux (GORD)
* renal failure
* severe cerebral palsy
* some enteropathies
* oesophageal strictures
* achalasia
* diabetes mellitus with gastroparesis
* surgical contra-indications
* Emergency cases
* patients that were already intubated

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Gastric residual volume by ultrasound after application of clear fluid fasting for 1 hour versus 2 hours prior to general anaesthesia | Prior to induction of general anaesthesia
  We use ultrasound to evaluate gastric volume We scanning distal parts of the stomach-antrum in a semi-sitting or RLD position.
  A linear high-frequency (e.g. 5-12 MHz) transducer can be used in leaner or paediatric patients or to obtain detailed images of the gastric wall(4-6mm).
  Antral cross sectional area(CSA) can be measured by using two perpendicular diameters and the formula of the area of an ellipse: CSA=(AP×CC×π)/4 (AP=antero-posterior diameter and CC=craniocaudal diameter)
  GV (ml)=27.0+14.6×right-latCSA-1.28×age(Perlas and colleagues formula)
  Total gastric residual volume is then divide by body weight to get ml/kg, the lower the value the better the outcome.
  Referance standard is gastric residual volume acquired through nasogastric suction using nasogastric tube.
  Result of >1.5ml/kg show that patient posed risk of aspiration, result of >1ml/kg is significantly increase in this study

SECONDARY OUTCOMES:
Anxiety level of patients by short version of(mYPAS)modified Yale Preoperative Anxiety Scale after application of clear fluid fasting for 1 hour versus 2 hours prior to paediatric general anaesthesia | Prior to induction of general anaesthesia and 1 hour post anaesthesia
  Total score from 22.916(minimum score= least anxiety level/total relaxation) to 100 (maximum score= maximum anxiety level/ panic attack)
  Total score is obtained from 4 subscale as describe below:
  A. Activity (1-4) B. Vocalizations(1-6) C. Emotional expressivity(1-4) D. State of apparent arousal (1-4) Total score: Divide each item rating by the highest possible rating (i.e., 6 for the "vocalizations" item and 4 for all other items), add all of the produced values, divide by 4, and multiply by 100
Parental satisfaction by questionnaires after application of clear fluid fasting for 1 hour versus 2 hours prior to paediatric general anaesthesia | 2 hours to 24 hours post anaesthesia
  Total score from 20(minimum score= not satisfy) to 100 (maximum score= highly satisfy) Total score is obtained from 11 answer to the 11 questions
  each of the answer will be score as: Strongly Agree(5 )- Agree(4 )- Neither Agree nor Disagree(3)- Disagree(2) -Strongly Disagree(1) except answers for questionnaire number 3,6,8 will be score as: Strongly Agree(1 )- Agree(2 )- Neither Agree nor Disagree(3)- Disagree(4) -Strongly Disagree(5) Total score calculation: Divide each item rating by 5, add all of the produced values, divide by 11, and multiply by 100

CONTACTS AND LOCATIONS:
Overall Officials: Ma Tai Jiun, Dr, Principal Investigator — University of Malaya; Ina Ismiarti binti Shariffuddin, Ass. Prof, Study Chair — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
The IPD will not be share because the IPD data is not particularly important in deciding the feasibility of 1 hour clear fluid fasting guideline.